CLINICAL TRIAL: NCT06437990
Title: Pilot Study of Arteriovenous Loop Graft for Free Functional Gracilis Transfer in Brachial Plexus Injured Patients With Insufficient Flow of Donor Artery
Brief Title: Arteriovenous Loop Graft for Free Functional Gracilis Transfer in Brachial Plexus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Panai Laohaprasitiporn, MD, Assistant Professor, Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 652/2556(EC4)
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Brachial Plexus Injury
Keywords: brachial plexus injury; brachial plexus palsy; free functional muscle transfer; arteriovenous loop graft; subclavian artery injury; axillary artery injury

STUDY DESIGN:
Intervention Model Description: Late-onset brachial plexus injury patient with concomitant subclavian or axillary artery injury
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arteriovenous loop graft (Experimental): A saphenous vein graft was used to create an arteriovenous loop from the common carotid artery to the external jugular vein, providing vascular supply for a free functional gracilis muscle flap in patients with late-onset brachial plexus injury.
  Interventions: Procedure: Arteriovenous loop graft

INTERVENTIONS:
Procedure: Arteriovenous loop graft — Using saphenous vein graft to create an arteriovenous loop from the common carotid artery to the external jugular vein, providing vascular supply for a free functional gracilis muscle flap in patients with late-onset brachial plexus injury with concomitant subclavian or axillary artery injury.
  Other Names: AV loop graft

SUMMARY:
Free functional muscle transfer (FFMT) using the gracilis muscle as a donor muscle has become a standard treatment for reconstructing late-onset brachial plexus injuries. Successful implementation of this procedure relies on the availability of functional donor vessels in the injured limb to supply the muscle flap. However, some brachial plexus injuries are accompanied by subclavian or axillary artery injuries, which compromise the viability of the muscle flap due to insufficient vascular supply. To address this, arteriovenous (AV) loop grafts have been employed to extend donor vessels to the flap and have been utilized in various body regions, including the upper extremity. Despite their widespread use, AV loop grafts have not been previously utilized in FFMT for late-onset brachial plexus injuries with concurrent subclavian or axillary artery injuries. This study aimed to assess the feasibility of this surgical approach and report the long-term outcomes of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or more than 20 years old
* Patients with brachial plexus injury with depletion of blood flow to the injured limb which confirmed by abnormal computed tomography arteriogram

Exclusion Criteria:

* Patients who had sufficient thoraco-acromial or thoraco-dorsal artery blood flow for standard free functional muscle transfer operation without the need of an AV loop graft

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Viability of the flap | 1 month
  Survival of the flap after the surgery

SECONDARY OUTCOMES:
Motor power | 12 months, 18 months
  Medical Research Council (MRC) grading for motor power assessment
Complications | 1 month
  Bleeding, infection, blood transfusion, stroke, embolism, thrombosis
Operative time | 1 month
  Total operative time including flap revision surgery or other related complications

CONTACTS AND LOCATIONS:
Overall Officials: Panai Laohaprasitiporn, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Limthongthang R, Wongtrakul S, Laohaprasitiporn P, Monteerarat Y, Vathana T. Free Functional Muscle Transfer in Brachial Plexus Injury Patients With Subclavian Artery Injury Using Arteriovenous Loop Grafts. Microsurgery. 2025 Jan;45(1):e70020. doi: 10.1002/micr.70020. PMID 39775958